CLINICAL TRIAL: NCT00876954
Title: Preoperative Whole-Body Hyperthermia in Patients Undergoing Major Abdominal Cancer Surgery: A Randomized Pilot Study
Brief Title: Preoperative Hyperthermia in Major Abdominal Surgery Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Braun Stiftung (Unknown)
Responsible Party: Principal Investigator, Oliver Kimberger, Assoc.Prof.PD Dr. MSc, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PreopHypertherm1
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Diathermy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Warming without increase in core temperature
  Interventions: Procedure: Normothermia
- Hyperthermia (Active Comparator): Hyperthermia for 2,5 hours (39 °C core temperature)
  Interventions: Procedure: Hyperthermia

INTERVENTIONS:
Procedure: Normothermia — Warming without increase in core temperature
  Arms: Placebo
Procedure: Hyperthermia — Core hyperthermia (39 °C) for 2,5 hours
  Arms: Hyperthermia

SUMMARY:
The investigators hypothesize that preoperative hyperthermia improves postoperative complications and compare a placebo group with standard thermoregulatory management (normothermia) to a treatment group receiving 2,5 hours of hyperthermia (38.5-39.5 °C core temperature) in a randomized, single blinded, controlled trial.

DETAILED DESCRIPTION:
The investigators hypothesize that preoperative hyperthermia improves postoperative complications and compare a placebo group with standard thermoregulatory management (normothermia) to a treatment group receiving 2,5 hours of hyperthermia (38.5-39.5 °C core temperature) in a randomized, single blinded, controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, age 18 - 75
* Open abdominal, curative cancer surgery > 2 h

Exclusion Criteria:

* Pregnancy
* Chronic cortisone treatment
* Ongoing chemotherapy
* Acute infections, septic surgery
* Palliative surgery (e.g. debulking only)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-04; Primary Completion 2010-10 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Immune Status | 24 hours after surgery
  LPS induced TNF-alpha

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Kimberger, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Oliver Kimberger M.D., Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided
on request